CLINICAL TRIAL: NCT03379155
Title: ZIEL - Zurück Ins Eigene Leben - Internet-based Self-help for Negative Life Events
Brief Title: Internet-based Self-help for Negative Life Events
Acronym: ZIEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZIEL
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Adjustment Disorders
MeSH Terms: conditions — Adjustment Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial design, comparing to a waitling list
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (Experimental): Internet-based self-help
  Interventions: Other: Internet-based self-help program
- Waiting List Group (No Intervention)

INTERVENTIONS:
Other: Internet-based self-help program — The intervention provided is based on the principles of cognitive behavioral therapy (CBT) (Bachem & Maercker, 2013). The manual integrates a variety of approaches validated as treatments for PTSD, anxiety disorders, or depression; the selection focuses on exercises which are intended to target the main symptoms of AjD, namely preoccupations (e.g. constant rumination, excessive worry about the stressor) and failure to adapt (e.g. sleep disturbance, difficulties concentrating, loss of interest in previously enjoyable activities).
  Arms: Active Group

SUMMARY:
The purpose of the study is to investigate the efficacy of an internet-based self-help intervention for dealing with stressful life events.

DETAILED DESCRIPTION:
The purpose of the study is to investigate the efficacy of an internet-based self-help intervention for dealing with stressful life events compared to a waiting list, in a randomized controlled trial design. Assessments are at baseline, 4-week and 3 months post-randomization. After 4 weeks, participants in the waiting control group get also access to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Negative life event in a period between two weeks and two years before the study
* Internet account
* Sufficient German language skills
* Informed consent

Exclusion Criteria:

* Persons with moderate or severe depressive symptoms
* Acute suicidality
* Psychotic disorder, bipolar disorder
* Severe, acute mental or physical disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Adjustment Disorder - New Module 20 (ADNM-20) | 4-week
  The ADNM-20 is a self-report assessment for adjustment disorder. It is aimed at adults who feel burdened by a critical life event.
  The ADNM-20 consists of two parts: an event list for recording stress and an item list for recording the resulting symptoms. In the event list, all burdens during the last two years are recorded and the subjectively highest burdens are named. On the basis of the item list, preoccupations and mismatch, the main symptom groups of the adaptation disorder according to ICD-11, as well as the concomitant symptoms of avoidance, depressiveness, anxiety, impulse control problems and functional impairment are recorded.
  The scale ranges from 0 (no stress) to 80 (high exposure).

SECONDARY OUTCOMES:
Brief Symptom Inventory - Short Version (BSI-18) | 4-week
  The short version of the Brief Symptom Inventory (BSI-18) is an easily applicable, reliable and valid self-report measure in wide international use. It assesses the syndromes of somatisation, depression and anxiety by means of 6 items each.
  The global factor ranges from 0 (no symptoms) to 72 (high symptomatic burden).
Beck Depression Inventory (BDI) | 4-week
  The BDI is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression.
  The score ranges from 0 (no symptoms) to 63 (severe depression).
Short Form 12-Item Survey (SF-12) | 4-week
  The SF-12 consists of 12 questions and is a general health questionnaire that provides information on the patient's state of health in more than 8 different dimensions.
  Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Sense of Coherence Questionaire Revised (SOC-R) | 4-week
  The SOC-R is a new conceptualization and operationalization of the resilience indicator SOC.
  The total score ranges from 13 (low) to 65 (high SOC).
Questionnaire for measuring patient satisfaction (ZUF-8) | 4-week
  The ZUF-8 is a self-assessment tool to assess the patient's satisfaction with regard to aspects of the clinic and treatment.
  The scale ranges from 8 (bad) to 32 (good satisfaction).
Credibility/Expectancy Questionaire (CEQ) | 4-week
  The CEQ is a scale for measuring treatment expectancy and rationale credibility for use in clinical outcome studies.
  The CEQ utilizes two scales during the administration (1-9, and 0-100%).
System Usability Scale (SUS) | 4-week
  The System Usability Scale (SUS) is a simple and technology-independent questionnaire to evaluate the usability of a system.
  The score ranges from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Maercker, Prof., Study Chair — Universität Zürich
Locations (2):
- Switzerland (2):
  - University of Bern, Bern
  - Universität Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No